CLINICAL TRIAL: NCT05983081
Title: Efficacy of Intra-articular Hyaluronate Injection for Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chih-Ya Chang, Tri-Service General Hospital, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSGH
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Adhesive Capsulitis
Keywords: frozen shoulder; hyaluronic acid
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: group A: intra-articular glenohumeral joint injections with HA, 60mg, once per week for 3 consecutive weeks.
  group B: physical therapy
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection Treatment (Experimental): A- Experimental Group: Intra-articular Hyaluronic Acid Injection Treatment Regimen Patients in the experimental group received ultrasound-guided intra-articular injections of hyaluronic acid (Artibest, 60 mg/3 ml, 2%, manufactured by Kang Stem Biotech, Taiwan) into the affected shoulder joint. The injections were administered once a week for three consecutive weeks, totaling three injections per patient. The subjects were evaluated for shoulder function using the Shoulder Pain and Disability Index (SPADI) and Range of Motion (ROM) assessment at the following time points: before the treatment, 4 weeks after the treatment, 6 weeks after the treatment, and 8 weeks after the treatment.
  Interventions: Procedure: Injection Treatment
- Physical Therapy (No Intervention): B- Control Group: Physical Therapy Patients in the control group underwent a 6-week physical therapy program, consisting of two sessions per week, with each session lasting approximately 30 minutes. The physical therapy program was conducted under the guidance and supervision of a physical therapist and included joint exercises, stretching, and muscle strengthening exercises.

INTERVENTIONS:
Procedure: Injection Treatment — Physical Therapy
  Arms: Injection Treatment

SUMMARY:
Objective: To evaluate the efficacy of intra-articular hyaluronic acid (HA) injections for the treatment of adhesive capsulitis (AC) of the shoulder.

Design: Prospective, case- controlled trial. Setting: Rehabilitation department of a medical center hospital. Participants: Patients (30) with AC Interventions: The patients received intra-articular glenohumeral joint injections of HA, 60mg, once per week for 3 consecutive weeks.

Main Outcome Measures: Active and passive range of motion (ROM) of the affected shoulder; Shoulder pain and disability were measured using 2 questionnaires: the SPADI. The patients were evaluated before treatment and were reevaluated 4, 6, 8, 12 weeks after the beginning of the treatment.

ELIGIBILITY:
Inclusion Criteria:

A. Patients diagnosed with frozen shoulder by a clinical physician based on the patient's medical history, physical examination, X-ray, and ultrasound or magnetic resonance imaging reports.

B. Clinical course: Patients must have a pain score of less than 3, no nighttime shoulder pain, and be in the post-freezing stage, primarily presenting restricted shoulder joint range of motion.

C. The affected shoulder joint must have at least two angles of shoulder joint movement reduced by at least 30% compared to the healthy side: shoulder flexion, abduction, and external rotation, or a single affected side abduction angle reduced by 50% relative to the healthy side.

D. Age between 40 to 70 years old.

-

Exclusion Criteria:

A. full-thickness tear or massive tear of the rotator cuff tendons or calcific tendinitis.

B. Presence of systemic rheumatic disease. C. History of shoulder fracture or previous shoulder surgery. D. Received shoulder injections for treatment within the last 3 months. E. Acute cervical nerve root compression. F. Current pregnancy or lactation. G. Patients with shoulder instability or cancer. H. Patients with cognitive impairment, unable to follow simple instructions, or unable to comply with the study procedures.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index | before the treatment, 4 weeks after the treatment, 6 weeks after the treatment, and 8 weeks after the treatment.
  The SPADI consists of two subscales, pain, and disability, comprising a total of 13 items. Each item is rated on a scale from 0 (no pain/disability) to 10 (most severe pain/disability). Higher scores indicate greater functional impairment. The total score on the SPADI is used to determine the percentage of functional disability

SECONDARY OUTCOMES:
Range of Motion | before the treatment, 4 weeks after the treatment, 6 weeks after the treatment, and 8 weeks after the treatment.
  The ROM is assessed using a standardized goniometer in the standard position to measure the angles of shoulder joint movement on the affected side. It includes flexion, extension, abduction, external rotation, and internal rotation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Alberta, Taiwan

IPD SHARING:
Plan to Share IPD: No